CLINICAL TRIAL: NCT06790537
Title: Efficacy of Pregabalin for Diabetic Pruritus - A Randomized Controlled Study.
Acronym: PREDICT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PREDICT
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Pruritus; Efficacy of Pregabalin in Controlling Diabetic Pruritus Severity
Keywords: Efficacy of pregabalin for control of generalised pruritus in Diabetic patients
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Pregabalin with emollient group. Pregabalin 75 mg one dose at night plus emollient application in the morning after bathing.
  Interventions: Drug: Pregabalin 75 mg
- placebo arm (Placebo Comparator): Placebo pill identical in appearance to the pregabalin capsule and standard treatment with emollient application locally on the areas of itching .
  Interventions: Other: Placebo Oral Capsule

INTERVENTIONS:
Drug: Pregabalin 75 mg — 75 mg of pregabalin will be given at night for the intervention group along with emollient local application
  Arms: Intervention group
Other: Placebo Oral Capsule — placebo capsule will be identical in appearance to the pregabalin capsule. it will be given at the same time of the day like pregabalin. same Emollient which is used in the Intervention arm will be applied locally on the areas of itching, morning after bathing .
  Arms: placebo arm

SUMMARY:
Brief Summary:

The goal of this randomized controlled study is to learn if pregabalin combined with emollients can reduce pruritus (itching) in people with Type 2 Diabetes Mellitus. The main questions it aims to answer are:

Does pregabalin combined with emollients reduce pruritus severity compared to a placebo combined with emollients? What is the impact of pregabalin on the quality of life of participants suffering from diabetic pruritus? we will compare pregabalin plus emollient to a placebo plus emollient to see if pregabalin works better for reducing pruritus.

Participants will:

Receive either pregabalin 75 mg daily along with emollient therapy or a placebo along with emollient therapy.

Visit the clinic at weeks 4, 8, and 12 for follow-up assessments, including:

Pruritus severity using the Visual Analog Scale (VAS) and 5-D Itch Scale. Patient Global Impression of Change (PGIC) to measure overall improvement. This study will help determine if pregabalin, a drug used for neuropathic pain, can be an effective treatment for pruritus in people with diabetes.

DETAILED DESCRIPTION:
Introduction Pruritus, commonly referred to as itching, is a common symptom experienced by patients with diabetes mellitus (DM). It is associated with both physical discomfort and significant psychological distress, affecting the overall quality of life (QoL). While acute pruritus may act as a protective response to harmful stimuli, chronic pruritus lasting for more than six weeks often signals an underlying pathology. In diabetic patients, pruritus can result from a combination of metabolic, neuropathic, and dermatological factors, leading to persistent symptoms. Despite its high prevalence, effective treatments for diabetic pruritus remain limited.

Pruritus in diabetes mellitus is complex, often resulting from diabetic neuropathy, skin barrier dysfunction (xerosis), and oxidative stress. Although treatments like emollients and antihistamines are used, their effectiveness is often suboptimal, particularly since diabetic pruritus is primarily non-histaminergic in nature. Pregabalin, a medication commonly used for neuropathic pain, has shown promise in treating neuropathic pruritus. Given the neuropathic component of diabetic pruritus, pregabalin may provide an effective treatment option when combined with emollients to address skin dryness.

Rationale for the Study Diabetic pruritus presents a significant challenge due to its multifactorial nature. While various treatments such as topical agents and antihistamines are used, they do not effectively address the underlying neuropathic component of pruritus in diabetic patients. Pregabalin, by modulating calcium channels and reducing neuronal excitability, has demonstrated efficacy in treating neuropathic pruritus in conditions such as uremic pruritus. Considering that diabetic pruritus shares similar neuropathic mechanisms, pregabalin could represent a valuable treatment option for reducing pruritus severity.

Additionally, xerosis (dry skin) is a common issue in diabetic patients and contributes significantly to pruritus. Emollient therapy helps restore moisture to the skin, addressing this underlying factor. The combination of pregabalin and emollient therapy may therefore provide a synergistic effect, reducing pruritus severity and improving the QoL of diabetic patients.

Aim:

To assess the efficacy of pregabalin combined with emollient therapy in reducing the severity of pruritus in patients with Type 2 Diabetes Mellitus (T2DM), compared to a placebo combined with emollient therapy.

Primary and Secondary objectives:

Primary Objective:

VAS Score: The mean change in VAS scores from baseline to week 12 between the pregabalin and placebo groups. The VAS measures pruritus severity, where patients rate their itch intensity from 0 (no itch) to 10 (worst imaginable itch).

Secondary Objective :

Proportion of participants achieving a minimum 3-point reduction in VAS scores at week 12.

Mean change in VAS scores at weeks 4 and 8. 5-D Itch Scale: A multidimensional scale measuring pruritus across five domains: duration, degree, direction, disability, and distribution.

PGIC Scores: The Patient Global Impression of Change scale is a subjective measure of the patient's overall perception of improvement, assessed at weeks 4, 8, and 12.

Safety Profile: Incidence and severity of adverse events (AEs) during the study period.

Discontinuation Rates: Rates of participant withdrawal due to adverse events in both treatment groups.

Inclusion Criteria:

Adults aged >18 years with Type 2 Diabetes Mellitus. HbA1c <10% with stable medication for at least 1 month before enrollment. Chronic pruritus lasting for six weeks or longer. Generalized or localized pruritus affecting more than one major body area as per the 5-D Itch Scale distribution.

Baseline VAS score ≥ 5.

Exclusion Criteria:

Type 1 Diabetes Mellitus, gestational diabetes, pregnant or breastfeeding women.

Pruritus duration of less than six weeks. Pruritus associated with conditions such as uremia (CKD stage IV/V), cholestasis, viral hepatitis, HIV, uncontrolled hypothyroidism, uncontrolled hyperthyroidism, and others.

Pruritus due to primary dermatological disorders (e.g., eczema, psoriasis, lichen planus).

Recent use of systemic treatments affecting pruritus, including gabapentins, tricyclic antidepressants, antihistamines, corticosteroids, or calcineurin inhibitors (within 2 weeks before study initiation).

Known hypersensitivity to pregabalin or emollients. Severe psychiatric disorders that may interfere with the evaluation of pruritus or adherence to the study.

Immunocompromised patients (e.g., post-transplant, immunosuppressive therapy). Methodology

Study Design:

This is a double-blind, randomized controlled trial (RCT). Both participants and researchers will be unaware of the treatment allocation, ensuring unbiased results.

Study Population:

The study will include adults aged 18 and above, diagnosed with Type 2 Diabetes Mellitus, who are experiencing chronic pruritus for at least six weeks.

Intervention:

Group A (Intervention): Pregabalin 75 mg daily at night + emollient therapy. Group B (Control): Placebo (identical to pregabalin) + emollient therapy.

Randomization:

Participants will be randomly assigned to one of the two treatment groups using a computer-generated randomization schedule to maintain allocation concealment.

Follow-up and Assessments:

Participants will attend follow-up visits at weeks 4, 8, and 12 for:

Pruritus severity assessment using VAS and 5-D Itch Scale. PGIC evaluation to assess subjective improvement. Safety monitoring for adverse events.

Statistical Analysis:

The primary endpoint is the change in VAS scores from baseline to week 12. Secondary endpoints include changes in the 5-D Itch Scale, PGIC scores, and safety assessments.

Appropriate statistical tests (e.g., t-tests, chi-square tests) will be used for comparisons between groups.

Ethical Considerations This study will be conducted in accordance with ethical guidelines provided by the Declaration of Helsinki and Good Clinical Practice (GCP). Ethical approval will be obtained from the Institutional Ethics Committee (IEC) of PGIMER, Chandigarh, and informed consent will be obtained from all participants.

Conclusion This study aims to evaluate the efficacy of pregabalin in treating diabetic pruritus, a common and troublesome symptom for diabetic patients. The combination of pregabalin and emollients may provide a novel, effective approach for managing pruritus and improving the quality of life for those affected.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>18 years) with Type 2 Diabetes Mellitus
2. HbA1c <10% and on stable medication for at least 1 month before enrolment.
3. Presence of chronic pruritus (lasting for six weeks or longer) [2].
4. Generalized or localised pruritus affecting more than one major body area*
5. Baseline VAS score of ≥5 $ *Pruritus including Generalized or localized pruritus as long as it involves two or more areas as per the 5D Itch Scale distribution [Head/scalp, face, chest, abdomen, back, buttocks, thighs, lower legs, feet/toes, arms, palms, hands/fingers, groin, and clothing contact points (waistbands/undergarments).

$ Baseline VAS score of ≥5 is included to ensure sufficient severity of pruritus for measurable improvement.

Exclusion Criteria:

1. Types of Diabetes:

   o Gestational Diabetes, pregnant and breastfeeding women with T2DM, Type 1 DM.
2. Pruritus Duration and Causes:

   * Pruritus of less than six weeks' duration.
   * Pruritus associated with systemic conditions such as uraemia (CKD stage IV/V), cholestatic liver diseases, viral hepatitis, HIV infection, uncontrolled hypothyroidism* or hyperthyroidism^, myeloproliferative disorders, Chronic venous insufficiency in legs or Postherpetic pruritus.

     *Uncontrolled hypothyroidism - T3 / T4 below the upper limit of normal.

     ^Uncontrolled hyperthyroidism- T3/T4 above the upper limit of normal.
   * Pruritus due to primary dermatological disorders presenting with skin lesions (e.g., atopic dermatitis, eczema, psoriasis, allergic contact dermatitis, urticarial disorders, lichen planus, prurigo nodularis, asteatotic dermatitis).
3. Use of Medications Affecting Pruritus:

   o Current or recent use (within 2 weeks before study initiation) of systemic treatments that may impact pruritus, including gabapentins (e.g., pregabalin, gabapentin), tricyclic antidepressants (TCA), antihistamines, corticosteroids, and calcineurin inhibitors.

   Rationale: Since these medications are commonly used for neuropathic pain or Pruritus which coexists with diabetic pruritus, their recent use may affect pruritus severity and treatment response. Patients using these drugs for neuropathic pain or other conditions should undergo a washout period of 2 weeks before study initiation.
4. Drug Hypersensitivity and Reactions:

   o Known allergies or hypersensitivity to pregabalin or emollient.
5. Psychiatric and Immunocompromised Status:

   * Severe psychiatric disorders that may interfere with the evaluation of pruritus or adherence to the study protocol.
   * Immunocompromised patients (e.g., post-transplant, immunosuppressive therapy). Pruritus due to Notalgia paresthetica or brachioradial pruritus, post burn pruritus, opioid-induced pruritus.
6. People with Substance abuse disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
• Mean change in VAS (Visual analogue scale)scores from baseline to week 12 between the two groups. | 12 weeks
  For all patients baseline VAS score will be assessed , then for both the intervention groups , follow up VAS scores will be noted at week 4, 8 and 12 weeks. Mean change in VAS scores in both the groups before and after the intervention will be the Primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ashu Rastogi, DM ENDOCRINOLOGY, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Department of Endocrinology , PGIMER, Chandigarh, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided